CLINICAL TRIAL: NCT03882463
Title: Interest of SmartGuard Technology (Predictive System for Stopping Insulin Before Hypoglycemia) in Children With Type 1 Diabetes Treated With Insulin Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO19026*
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- insulin pump function (Experimental): continuous glucose monitoring and then continuous glucose monitoring with the stop insulin pump function
  Interventions: Device: Continuous glucose monitoring with the stop insulin pump function

INTERVENTIONS:
Device: Continuous glucose monitoring with the stop insulin pump function — Children with type 1 diabetes using insulin pump and continuous glucose monitoring without the stop insulin pump functionare then using the predictive system for stopping before hypoglycaemia "medtronic Minimed with SmartGuard technology".

SUMMARY:
Management of children and adolescents with type 1 diabetes is essentially insulin therapy using insulin pump, allowing the improvement of the glycemic balance.

However, the risk of hypoglycaemia inherent to the treatment persists. Hypoglycemia is an acute complication in the management of diabetes. It can be manifested by warning signs (tremors, sweats, feelings of hunger ...) but also occur during sleep and be ignored. It can be responsible for asthenia, difficulty concentrating and attention and memory problems.

In order to decrease time spent in hypoglycemia, insulin pump therapy can be coupled with a continuous glucose measurement system with a stop insulin pump function in case of hypoglycemia.

The aim of the study is to evaluate efficacy of the predictive system for stopping before hypoglycaemia "medtronic Minimed with SmartGuard technology" in type 1 diabetic children, especially on the time spent in hypoglycemia .

DETAILED DESCRIPTION:
Management of children and adolescents with type 1 diabetes is essentially insulin therapy using insulin pump, allowing the improvement of the glycemic balance.

However, the risk of hypoglycaemia inherent to the treatment persists. Hypoglycemia is an acute complication in the management of diabetes. It can be manifested by warning signs (tremors, sweats, feelings of hunger ...) but also occur during sleep and be ignored. It can be responsible for asthenia, difficulty concentrating and attention and memory problems.

In order to decrease time spent in hypoglycemia, insulin pump therapy can be coupled with a continuous glucose measurement system with a stop insulin pump function in case of hypoglycemia.

The aim of the study is to evaluate efficacy of the predictive system for stopping before hypoglycaemia "medtronic Minimed with SmartGuard technology" in type 1 diabetic children, especially on the time spent in hypoglycemia .

ELIGIBILITY:
inclusion criteria :

* children aged between 1 and 17 years
* type 1 diabetes
* Duration of type 1 diabetes > 1 year
* insulin pump therapy > 3 months

exclusion criteria :

* Other diseases predisposing to hypoglycemia
* Oral glycemic medications
* have used continuous glucose monitoring during the last 3 months
* HbA1c >10%

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time spent hypoglycemia | 1 month
  average daily time spent in hypoglycemia measured on a one-month data collection

SECONDARY OUTCOMES:
Number of hypoglycemia | 1 month
  Number of glycemia less than 0.70 g/l measured on a one-month data collection

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided